CLINICAL TRIAL: NCT05495945
Title: Ultrasonic Deep Brain Stimulation During Anesthetic Sedation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Zirui Huang, Research Assistant Professor, Anesthesiology and Research Fellow, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00213014; 2R01GM103894-10A1 (NIH)
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Mental Function
Keywords: Propofol; Anesthesia; Ultrasound; fMRI
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Dorsolateral prefrontal cortex (DLPFC) (Experimental)
  Interventions: Device: Low-intensity focused ultrasound pulsation (LIFUP); Combination Product: Functional Magnetic Resonance Imaging (fMRI) using Propofol
- Anterior insula cortex (AIC) (Experimental)
  Interventions: Device: Low-intensity focused ultrasound pulsation (LIFUP); Combination Product: Functional Magnetic Resonance Imaging (fMRI) using Propofol
- Central thalamus (CT) (Experimental)
  Interventions: Device: Low-intensity focused ultrasound pulsation (LIFUP); Combination Product: Functional Magnetic Resonance Imaging (fMRI) using Propofol
- Sham control (Active Comparator)
  Interventions: Combination Product: Functional Magnetic Resonance Imaging (fMRI) using Propofol

INTERVENTIONS:
Device: Low-intensity focused ultrasound pulsation (LIFUP) — LIFUP will be used to stimulate specific brain regions and assess their causal involvement in the control of conscious state and contents.
  Arms: Anterior insula cortex (AIC); Central thalamus (CT); Dorsolateral prefrontal cortex (DLPFC)
Combination Product: Functional Magnetic Resonance Imaging (fMRI) using Propofol — Propofol will be administered by intravenous infusion. All anesthesia equipment, supplies, and drugs will be provided by anesthesiologists from the University of Michigan Health System. The researchers will manually control the infusion of propofol to achieve target effect-site concentrations
  Other Names: Diprivan

SUMMARY:
The purpose of this study is to see if mental functions take place during different levels of anesthesia. The researchers expect to gain a deeper understanding of mental function during different levels of anesthesia, and to evaluate if the use of ultrasonic brain stimulation accelerates return to consciousness.

DETAILED DESCRIPTION:
The decision was made in 2023 to focus on the Central Thalmus arm only for this trial. Participants were only randomized to this arm.

ELIGIBILITY:
Inclusion Criteria:

* The participants will be right-handed adults
* Body mass index (BMI) less than 30.
* All subjects will be English speakers.

Exclusion Criteria:

* Participants will be excluded if they have any medical contraindication to MRI scanning
* Unable to undergo MRI scanning because of possible pregnancy or currently breastfeeding,
* BMI>30
* Metallic substances in the body, claustrophobia, anxiety, or cardiopulmonary disease;
* Intracranial structural abnormality on T1-weighted MRI scans.
* Potential subjects will be excluded if they have a history of allergy to propofol, eggs or egg products, soybean or soybean products,
* Neurological, cardiovascular, or pulmonary illness;
* Head injury with loss of consciousness;
* Learning disability or other developmental disorder; sleep apnea or any severe snoring history;
* Gastroesophageal reflux disease (GERD) or heartburn;
* Pancreatitis or a history of pancreatitis, or sensory/motor loss sufficient to interfere with performance of the study. Participants with tattoos in the head or neck region will be excluded from study; other tattoos are subject to determination by investigators based on their assessment regarding participant safety. To eliminate aspiration risk subjects will also be excluded if they have had recent food or liquid intake (within 8 hours). Subjects will be excluded if they have a history of drug use, have a positive drug screen, are unwilling to abstain from alcohol for 24 hours prior to dosing, or have a current history of nicotine use. Women will be required to take a pregnancy test prior to participation to ensure a negative result. The pre-scan drug screen and pregnancy test will be paid for by the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zirui Huang, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants were consented but did not receive sedation, as they were used as "dry runs" to test behavioral responses without sedation.
  1 participant was consented but was a screen fail, so was not randomized.
  Participants for this trial were only randomized to the central thalamus arm.
Period: Overall Study
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Anterior Insula Cortex (AIC) | Central Thalamus (CT) | Sham Control
Started | 0 | 0 | 8 | 0
Completed | 0 | 0 | 8 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 4 participants were consented but did not receive sedation, as they were used as "dry runs" to test behavioral responses without sedation.
  1 participant was consented but was a screen fail, so was not randomized. Participants for this trial were only randomized to the central thalamus arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Anterior Insula Cortex (AIC) | Central Thalamus (CT) | Sham Control | Total
Number analyzed (Participants) | 0 | 0 | 8 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] |  |  | 25.1 (6.6) |  | 25.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 7 |  | 7
  Male |  |  | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  | 0 |  | 0
  Not Hispanic or Latino |  |  | 8 |  | 8
  Unknown or Not Reported |  |  | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  | 0 |  | 0
  Asian |  |  | 1 |  | 1
  Native Hawaiian or Other Pacific Islander |  |  | 0 |  | 0
  Black or African American |  |  | 0 |  | 0
  White |  |  | 7 |  | 7
  More than one race |  |  | 0 |  | 0
  Unknown or Not Reported |  |  | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  |  | 8 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygen Level Dependent (BOLD) Response to Visual Stimuli
Description: BOLD signal was measured by Magnetic Resonance Imaging (MRI) scanning of the brain in response to a visual stimuli. This method reflected changes in oxygenation of blood in the brain during a scene-processing task.
Time Frame: Up to 90 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of BOLD signal
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Anterior Insula Cortex (AIC) | Central Thalamus (CT) | Sham Control
Number analyzed (Participants) | 0 | 0 | 8 | 0
percentage of BOLD signal
  Baseline |  |  | 0.56 (0.03) |
  Following Intervention |  |  | 0.51 (0.06) |
Statistical Analysis 1: Comparison: Central Thalamus (CT); Test type: Superiority; p = 0.62, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Perceptual Criterion Derived From the Signal Detection Theory (SDT)
Description: SDT was a means of measuring participants' ability to differentiate between information-bearing patterns and random patterns that distract from the information. Perceptual criterion measured a participant's tendency to say "yes" or "no" when the participant was unsure if a signal was present. Perceptual criterion was measured on a scale from -1.0 to 1.0, with a score of 0 indicating no bias towards "yes" or "no". Negative scores meant a bias towards "yes" (more likely to say a signal was present), while positive scores meant a bias towards "no" (more likely to say a signal was absent).
Time Frame: Up to 90 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Anterior Insula Cortex (AIC) | Central Thalamus (CT) | Sham Control
Number analyzed (Participants) | 0 | 0 | 8 | 0
score on a scale
  Baseline |  |  | 0.56 (0.89) |
  Following Intervention |  |  | 0.80 (1.05) |
Statistical Analysis 1: Comparison: Central Thalamus (CT); Test type: Superiority; p = 0.18, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Sensitivity Derived From the Signal Detection Theory (SDT)
Description: SDT was a means of measuring participants' ability to differentiate between information-bearing patterns and random patterns that distract from the information. Sensitivity measured a participant's ability to differentiate between real and scrambled images on a scale from 0.0 to 1.0, with higher scores indicating better accuracy in detecting a signal when it was present and lower scores indicating more missed signals. A score of 1.0 was perfect sensitivity (i.e., never missing a real signal).
Time Frame: Up to 90 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Anterior Insula Cortex (AIC) | Central Thalamus (CT) | Sham Control
Number analyzed (Participants) | 0 | 0 | 8 | 0
score on a scale
  Baseline |  |  | 0.72 (0.50) |
  Following Intervention |  |  | 0.39 (0.58) |
Statistical Analysis 1: Comparison: Central Thalamus (CT); Test type: Superiority; p = 0.20, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Grip Force
Description: Participants' grip force of hand squeezing on a rubber ball in response to instructions was measured.
Time Frame: Up to 90 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Anterior Insula Cortex (AIC) | Central Thalamus (CT) | Sham Control
Number analyzed (Participants) | 0 | 0 | 8 | 0
mmHg
  Baseline |  |  | 13.8 (5.3) |
  Following Intervention |  |  | 11.9 (3.8) |
Statistical Analysis 1: Comparison: Central Thalamus (CT); Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 24 hours
Description: Participants were only randomized to the Central Thalamus arm.
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Anterior Insula Cortex (AIC) | Central Thalamus (CT) | Sham Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/8 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/8 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 4/8 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dorsolateral Prefrontal Cortex (DLPFC) (N=0) | Anterior Insula Cortex (AIC) (N=0) | Central Thalamus (CT) (N=8) | Sham Control (N=0)
Moderate Fatigue (General disorders) | NA | NA | 1 | NA
Mild Episode of Apnea (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | NA
Mild Tenderness at IV site (Skin and subcutaneous tissue disorders) | NA | NA | 1 | NA
Mild Head Tenderness at Ultrasound Site (Skin and subcutaneous tissue disorders) | NA | NA | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT05495945/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT05495945/ICF_001.pdf